CLINICAL TRIAL: NCT04214197
Title: An Open Label, Photo Documentation Study of Crisaborole Ointment 2% in Mild to Moderate Atopic Dermatitis
Brief Title: Study of Crisaborole Ointment 2% in Mild to Moderate Atopic Dermatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Gideon Piers Smith, Associate Director, CURTIS, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002349
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crisaborole (Other): Crisaborole is a low molecular weight benzoxaborole PDE-4 inhibitor for the treatment of mild-to-moderate atopic dermatitis in adults and children 2 years and above. Crisaborole ointment 2% is topically applied as a thin layer twice daily for 4 weeks to all AD lesions.
  Interventions: Drug: Crisaborole 2% Top Oint

INTERVENTIONS:
Drug: Crisaborole 2% Top Oint — Crisaborole is a low molecular weight benzoxaborole PDE-4 inhibitor for the treatment of mild-to-moderate atopic dermatitis in adults and children 2 years and above. Crisaborole ointment 2% is topically applied as a thin layer twice daily for 4 weeks to all AD lesions.

SUMMARY:
The purpose of this study is to document the timing of improvement in atopic dermatitis symptoms and severity following the application of crisaborole ointment 2% in patients 2 years or older with mild to moderate atopic dermatitis. Crisaborole ointment 2% will be applied topically twice daily for four weeks and progress will be assessed by photography and patient-reports.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female aged at least 2 years of age.
2. Subject has confirmed clinical diagnosis of active atopic dermatitis (AD) according to the Hanifin and Rajka criteria.
3. AD diagnosed at least 6 months prior to the screening visit and severity of disease has been stable for the past month.
4. Subject has a BSA covered with atopic dermatitis of at least 1% (excluding face, scalp, genitals, groin area) [face, genitals and groin will not for be used photos]
5. Subject has a global ISGA of mild (2) or moderate (3) at the baseline visit.
6. Subject must be willing to avoid excessive exposure to natural or artificial ultraviolet radiation.
7. Women of childbearing potential who are heterosexually active must practice a highly effective method of birth control such as an oral, injected or implanted hormonal methods of contraception, intrauterine device (IUD), spermicidal condom, male partner sterilization (the vasectomized partner should be the sole partner for that subject) or true abstinence. If a female subject's childbearing potential changes after start of the study (e.g., a woman who is not heterosexually active becomes active, a premenarchal woman experiences menarche), she must begin practicing a highly effective method of birth control, as described above.
8. Women of childbearing potential must have a negative pregnancy test at the baseline visit.
9. Willingness to participate in medical photography with end use by Pfizer for publication and medical education purposes
10. Subject and/or parent/ legal guardian has voluntarily signed and dated an informed consent form and assent form, if applicable, approved by Partners Institutional Review Board (IRB) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study (including photography consent).

Exclusion Criteria:

1. Clinically significant medical disorder, condition, or disease including other dermatologic conditions that may interfere with study assessments and photographs.
2. Recent psychiatric condition (within the past year) or active suicidal ideation or behavior.
3. Unstable AD (not having stable severity over the past month).
4. Significant active infection requiring systemic antibiotics.
5. Treatment with topical corticosteroids or topical calcineurin inhibitors within 2 weeks of the baseline visit.
6. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, is likely to require immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon gamma, Janus kinase inhibitors, azathioprine, methotrexate, etc.) during the study.
7. Treatment with biologics within 5 half-lives (if known) or 16 weeks before the baseline visit, whichever is longer.
8. Subject with any planned surgical or medical procedure that would overlap with study participation from screening through end of study
9. Currently has a malignancy or has a history of malignancy within 5 years before screening (except for a nonmelanoma skin cancer that has been adequately treated).
10. Is pregnant, nursing, or planning a pregnancy (women).
11. Previous failure of efficacy following crisaborole use.
12. History of angioedema or anaphylaxis to topical products.
13. Known allergies, hypersensitivity, or intolerance to crisaborole or its components.
14. Participation in another clinical research study with an investigational drug within 4 weeks before randomization in this study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Time to success (in days) on ISGA | At days 1, 8,15, 21 and 29
  Time to success (in days) on ISGA (to clear or almost clear with at least a 2-grade improvement) for intensive group through study completion, an average of 4 weeks, will be summarized by 25th percentile, median, and corresponding 95% CIs via Kaplan-Meier method. Kaplan-Meier plot will be provided as well.
Time to success (by week) on ISGA | At days 1, 8,15, 21 and 29
  Time to success (by week) on ISGA (to clear or almost clear with at least a 2-grade improvement) for all subjects through study completion, an average of 4 weeks, will be summarized by 25th percentile, median, and corresponding 95% CI via Kaplan-Meier method. Kaplan-Meier plot will be provided as well. (pooled all subjects, at days 1, 8,15, 21 and 29)

CONTACTS AND LOCATIONS:
Locations (1):
- MGH Clinical Unit for Research Trials in Skin (CURTIS), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weidinger S, Novak N. Atopic dermatitis. Lancet. 2016 Mar 12;387(10023):1109-1122. doi: 10.1016/S0140-6736(15)00149-X. Epub 2015 Sep 13. PMID 26377142
- [Background] Richard MA, Corgibet F, Beylot-Barry M, Barbaud A, Bodemer C, Chaussade V, D'Incan M, Joly P, Leccia MT, Meurant JM, Petit A, Geffroy BR, Sei JF, Taieb C, Misery L, Ezzedine K. Sex- and age-adjusted prevalence estimates of five chronic inflammatory skin diseases in France: results of the << OBJECTIFS PEAU >> study. J Eur Acad Dermatol Venereol. 2018 Nov;32(11):1967-1971. doi: 10.1111/jdv.14959. Epub 2018 Jul 16. PMID 29569785
- [Background] Deckers IA, McLean S, Linssen S, Mommers M, van Schayck CP, Sheikh A. Investigating international time trends in the incidence and prevalence of atopic eczema 1990-2010: a systematic review of epidemiological studies. PLoS One. 2012;7(7):e39803. doi: 10.1371/journal.pone.0039803. Epub 2012 Jul 11. PMID 22808063
- [Background] Silverberg JI. Public Health Burden and Epidemiology of Atopic Dermatitis. Dermatol Clin. 2017 Jul;35(3):283-289. doi: 10.1016/j.det.2017.02.002. Epub 2017 Apr 22. PMID 28577797
- [Background] Siegfried EC, Jaworski JC, Hebert AA. Topical calcineurin inhibitors and lymphoma risk: evidence update with implications for daily practice. Am J Clin Dermatol. 2013 Jun;14(3):163-78. doi: 10.1007/s40257-013-0020-1. PMID 23703374
- [Background] Castellsague J, Kuiper JG, Pottegard A, Anveden Berglind I, Dedman D, Gutierrez L, Calingaert B, van Herk-Sukel MP, Hallas J, Sundstrom A, Gallagher AM, Kaye JA, Pardo C, Rothman KJ, Perez-Gutthann S. A cohort study on the risk of lymphoma and skin cancer in users of topical tacrolimus, pimecrolimus, and corticosteroids (Joint European Longitudinal Lymphoma and Skin Cancer Evaluation - JOELLE study). Clin Epidemiol. 2018 Mar 13;10:299-310. doi: 10.2147/CLEP.S146442. eCollection 2018. PMID 29559812
- [Background] Gantner F, Gotz C, Gekeler V, Schudt C, Wendel A, Hatzelmann A. Phosphodiesterase profile of human B lymphocytes from normal and atopic donors and the effects of PDE inhibition on B cell proliferation. Br J Pharmacol. 1998 Mar;123(6):1031-8. doi: 10.1038/sj.bjp.0701688. PMID 9559883
- [Background] Chan SC, Reifsnyder D, Beavo JA, Hanifin JM. Immunochemical characterization of the distinct monocyte cyclic AMP-phosphodiesterase from patients with atopic dermatitis. J Allergy Clin Immunol. 1993 Jun;91(6):1179-88. doi: 10.1016/0091-6749(93)90321-6. PMID 8389777
- [Background] Tom WL, Van Syoc M, Chanda S, Zane LT. Pharmacokinetic Profile, Safety, and Tolerability of Crisaborole Topical Ointment, 2% in Adolescents with Atopic Dermatitis: An Open-Label Phase 2a Study. Pediatr Dermatol. 2016 Mar-Apr;33(2):150-9. doi: 10.1111/pde.12780. Epub 2016 Jan 18. PMID 26777394
- [Background] Paller AS, Tom WL, Lebwohl MG, Blumenthal RL, Boguniewicz M, Call RS, Eichenfield LF, Forsha DW, Rees WC, Simpson EL, Spellman MC, Stein Gold LF, Zaenglein AL, Hughes MH, Zane LT, Hebert AA. Efficacy and safety of crisaborole ointment, a novel, nonsteroidal phosphodiesterase 4 (PDE4) inhibitor for the topical treatment of atopic dermatitis (AD) in children and adults. J Am Acad Dermatol. 2016 Sep;75(3):494-503.e6. doi: 10.1016/j.jaad.2016.05.046. Epub 2016 Jul 11. PMID 27417017
- [Background] Murrell DF, Gebauer K, Spelman L, Zane LT. Crisaborole Topical Ointment, 2% in Adults With Atopic Dermatitis: A Phase 2a, Vehicle-Controlled, Proof-of-Concept Study. J Drugs Dermatol. 2015 Oct;14(10):1108-12. PMID 26461821
- [Background] Defining a responder on the Peak Pruritus Numerical Rating Scale (NRS) in patients with moderate-to-severe atopic dermatitis: Detailed analysis from randomized trials of dupilumab. Journal of the American Academy of Dermatology. 2017;76(6):AB93.
- [Background] Yosipovitch G, Reaney M, Mastey V, Eckert L, Abbe A, Nelson L, Clark M, Williams N, Chen Z, Ardeleanu M, Akinlade B, Graham NMH, Pirozzi G, Staudinger H, Plaum S, Radin A, Gadkari A. Peak Pruritus Numerical Rating Scale: psychometric validation and responder definition for assessing itch in moderate-to-severe atopic dermatitis. Br J Dermatol. 2019 Oct;181(4):761-769. doi: 10.1111/bjd.17744. Epub 2019 May 1. PMID 30729499
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Olsen JR, Gallacher J, Finlay AY, Piguet V, Francis NA. Quality of life impact of childhood skin conditions measured using the Children's Dermatology Life Quality Index (CDLQI): a meta-analysis. Br J Dermatol. 2016 Apr;174(4):853-61. doi: 10.1111/bjd.14361. Epub 2016 Mar 6. PMID 26686685
- [Background] Mirfeizi M, Jafarabadi MA, Toorzani ZM, Mohammadi SM, Azad MD, Mohammadi AV, Teimori Z. Feasibility, reliability and validity of the Iranian version of the Diabetes Quality of Life Brief Clinical Inventory (IDQOL-BCI). Diabetes Res Clin Pract. 2012 May;96(2):237-47. doi: 10.1016/j.diabres.2011.12.030. Epub 2012 Feb 1. PMID 22306060
- See also: MGH Dermatology — https://www.massgeneral.org/Dermatology/